CLINICAL TRIAL: NCT05788471
Title: Effect of Neurodynamic Mobilization on Median Nerve Conduction Velocity in Carpal Tunnel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Raghda Ahmed Mohammed Ebrahim, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Raghda Ahmed_PhD
Record Dates: First submitted 2023-03-15; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Median Nerve Entrapment; Carpal Tunnel Syndrome
MeSH Terms: conditions — Median Neuropathy; Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment group (Active Comparator): Twenty patients will receive conventional treatment in the form of superficial heat, ultrasound with freq of 1 MHz, pulsed mode 1:4 for 5 min and stretching exercise to lumbrical muscles of the hand.
  Interventions: Other: conventional Treatment
- Neurodynamic mobilization therapy group (Experimental): Twenty patients will receive neurodynamic mobilization therapy (upper limb tension test 1) in addition to conventional treatment.
  Interventions: Other: conventional Treatment; Other: Neurodynamic mobilization

INTERVENTIONS:
Other: conventional Treatment — It consists of Superficial heat, Ultrasound therapy and stretching exercise to lumbrical muscles of the hand.
Other: Neurodynamic mobilization — It is the mobilisation of the nervous system as an approach to physical treatment of pain. The treatment and or assessment relies on influencing pain physiology via the mechanical treatment of neural tissues and non-neural structures surrounding the nervous system.
  Arms: Neurodynamic mobilization therapy group

SUMMARY:
The purpose of this study is to examine:

1. The effect of neurodynamic mobilization on the sensory and motor median nerve conduction velocity in carpal tunnel syndrome.
2. The effect of neurodynamic mobilization on the wrist pain in carpal tunnel syndrome.
3. The effect of neurodynamic mobilization on the hand function in carpal tunnel syndrome.

DETAILED DESCRIPTION:
The findings of this study will provide physiotherapists with information to know if neurodynamic mobilization techniques is effective on median nerve conduction velocity in carpal tunnel syndrome also this will improve our body of knowledge about the best modalities for treating carpal tunnel syndrome. The finding of this study may help carpal tunnel syndrome patients to avoid the exposing to complications as a result of compression of median nerve in carpal tunnel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Forty carpal tunnel syndrome patients.
* All participants referred from a physician.
* Their ages range from 20-50 years old.
* Both genders will participate in the study.
* Their BMI ranges between 18.5-24.9kg/m2.
* All participants have carpal tunnel syndrome at least in one hand.
* All participants suffering from mild to moderate carpal tunnel syndrome.

Exclusion Criteria:

* Previous or current disease or trauma that might affect one or both upper limbs.
* Metabolic diseases that might associated with entrapment neuropathy such as diabetes mellitus, thyroid diseases, and autoimmune diseases.
* Pregnant women.
* Participants with congenital hand deformities.
* History of hand surgery.
* Sever cases of carpal tunnel syndrome that suffering from weakness of hand grip and atrophy of thenar muscle.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Assessing the change in nerve conduction velocity of the median nerve. | at baseline and after 4 weeks of intervention
  By using Electromyography apparatus measuring nerve conduction velocity of the median nerve. (motor and sensory in m/s)
Assessing the change in wrist joint pain | at baseline and after 4 weeks of intervention
  By using Pressure pain threshold (PPT) is defined as the minimal amount of pressure that produces pain. A simple handheld pressure algometer (PA) with a spring is commonly used, although more sophisticated electrical devices with a strain or pneumatic pressure gauge have been developed. They hold the peak force or pressure (kp (kilopond) = 10 N, Newton = 100 kPa (kilopascal)) until tared, and some may also be connected to a computer and thus have continuous output. PPT measured with a probe 1.6 mm in diameter or larger reflects the tenderness of deep tissues as anesthesia of skin only affects the results of smaller probes.
Assessing the change in functional activity of the hand | at baseline and after 4 weeks of intervention
  By using Modified DASH questionnaire will be used for functional activity of the hand. The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a 30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities. This questionnaire is a self-report questionnaire that patients can rate difficulty and interference with daily life on a 5 point Likert scale. The QuickDASH tool uses a 5-point Likert scale from which the patient can select an appropriate number corresponding to his/her severity/function level.

CONTACTS AND LOCATIONS:
Overall Officials: Raghda Ahmed, Principal Investigator — Cairo University
Locations (1):
- Outpatient clinic faculty of physica therapy cairo university, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Undecided